CLINICAL TRIAL: NCT03060200
Title: Reducing Depressive Symptomatology With a Smartphone App: A Protocol for a Randomized, Placebo-Controlled Clinical Trial
Brief Title: Reducing Depressive Symptomatology With a Smartphone App
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Babes-Bolyai University (Other)
Collaborators: Norwegian University of Science and Technology (Other); CheckWare AS (Unknown)
Responsible Party: Principal Investigator, Cezar Giosan, PhD, PhD, Babes-Bolyai University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EEA-JRP-RO-NO-2013-1-0358/2
Record Dates: First submitted 2017-02-01; First posted 2017-02-23 (Actual); Last update posted 2019-07-16 (Actual); Status verified 2019-07

CONDITIONS: Moderate Depression
Keywords: depression; treatment; CBT; online; app
MeSH Terms: conditions — Depression; Alzheimer Disease

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Active intervention (Experimental): Self-administered online CBT plus therapist check in. Moderately depressed participants will be testing a depression app, employing a self administered plus therapist check in, online CBT intervention, for 6 weeks.
  Interventions: Other: Self-administered online CBT plus therapist check in
- Waiting list (No Intervention): Moderately depressed participants will be put on a wait list for 6 weeks, after which access to the depression app will be given.
- Placebo (Placebo Comparator): Sham self-administered online CBT plus therapist check in. Moderately depressed participants will be using a depression app - the same platform and largely in the same format as the tested app, employing a self administered plus therapist check in, online sham intervention, for 6 weeks. The intervention will include the same sections and features as the original app, except for the complete exercises and behavioral activation sections. In addition, the psychoeducation section, although mirroring the structure of the corresponding section in the original app, will include different content, elaborating on common sense information on psychological well being.
  Interventions: Other: Sham self-administered online CBT plus therapist check in

INTERVENTIONS:
Other: Self-administered online CBT plus therapist check in — The app being tested is comprised of courses, exercises and a behavioural activation component. Courses represent the psycho-educational background of the program, comprising topics such as: information on depression, what is CBT, healthy/unhealthy negative emotions, rational/irrational thoughts, behaviour, social support, relaxation techniques, sleep hygiene, relapse prevention, treatment adherence, and suicide prevention plan. Exercises use the information presented in the courses and follow the structure of a regular therapy session/ therapeutic homework. The following exercises are included in the app: Emotional Pulse, Find Irrational Thoughts, and Change Irrational Thoughts. The behavioural activation component consists in two main exercises: My goals and My Activities.
  Arms: Active intervention
Other: Sham self-administered online CBT plus therapist check in — The active placebo intervention will be delivered via the same platform and largely in the same format as the tested app: it will include the same sections and features as the original app, except for the complete exercises. In addition, the psychoeducation section, although mirroring the structure of the corresponding section in the original app, will include different content, elaborating on common sense psychological well being aspects.
  Arms: Placebo

SUMMARY:
The aim of this study is to test a newly developed app, firmly grounded in Cognitive Behavioural Therapy (CBT) theory of depression, to determine primarily if this app is clinically useful in decreasing moderate depressive symptoms when compared with an active placebo. Additionally, we are interested in the app's potential to contribute to the reduction of general negative affect, increasing positive affect, and boosting satisfaction with life. Last, but not least, we aim to verify if the usage of the tested app can modify depressogenic cognitions.

DETAILED DESCRIPTION:
Trial design This study is a randomized, placebo-controlled trial, examining the effects of a CBT intervention in reducing depressive symptomatology for people with moderate symptoms. Participants are randomly assigned to one of the 3 arms of the trial: (1) CBT intervention; (2) placebo intervention (PI); and (3) delayed intervention (wait-list; WL). Major assessments are at baseline, post-treatment, and follow-up 12 weeks later. Participants randomized to the PI and WL trial arms are offered access to the online app upon completion of the study. Participants are blinded to hypotheses and the nature of the placebo intervention, but they are informed they have a 1 in 3 chance of being assigned to the placebo intervention.

Participant timeline Potential participants will be assessed for eligibility through an initial assessment of depressive symptoms. The initial assessment phase consists of administration of the Patient Health Questionnaire-9 (PHQ-9) and a short screening telephone interview. Applicants who do not meet the inclusion criteria are informed via e-mail. They are given a summary score and interpretation for their PHQ-9 score and they are encouraged to discuss their problems with a professional, if necessary. Information on how to reach one - a clinical psychologist or psychotherapist - is also provided. Subsequent assessments consist of all the instruments presented in the Outcome measures section. After the initial assessment, the participants meeting inclusion criteria will be randomly assigned to one of the three conditions: active intervention condition (Group 1), the placebo intervention (Group 2), and the delayed-intervention condition (wait-list) (Group 3).

The participants in the active intervention and active placebo conditions are assessed at pre-intervention (Time 1 - baseline), at mid-intervention (Time 2 - 3 weeks after baseline), at post-intervention (Time 3 - 6 weeks after baseline), and at 3-months post-intervention (Time 4). The participants in the delayed-intervention condition are assessed before the waiting period (Time 1 - baseline), at mid-waiting period (Time 2 - 3 weeks after baseline), and at post-waiting period (Time 3 - 6 weeks after baseline).

Participants assigned to the active intervention condition will be given access to the online application along with explicit instructions regarding the use of all of its sections. Participants will be given 6 weeks to complete the intervention, during which time weekly messages will be sent out to them. Messages include regular assignments designed for a complete and thorough use of the application's courses and exercises, and encourage the review of materials whenever possible. However, participants are free to use the application at their own pace.

Similarly, the participants in the active placebo condition will be given given access to a sham version of the app. During the 6-week intervention period they will be exposed to the same amount of online (i.e., in app messages) and therapist communication as the active intervention participants.

After each week, participants' application use is evaluated (see the Application Use Scale described above). Similarly, after each week of using the application, the participants are required to complete the Center for Epidemiologic Studies Depression Scale-Revised (CESD-R), for close monitoring of their depressive symptomatology and individualized feedback on their emotional state.

Participants in the delayed intervention condition are placed on a wait-list for 6 weeks, after which they are given access to the app.

Sample size A total number of 165 participants with moderate depressive symptomatology was estimated based on previous studies on the efficacy of mobile phone applications for depression that reported small to moderate between group effect sizes. An a priori sample size calculation was conducted with G*Power 3.1.9.2 for ANOVA (Repeated measures, between factors), assuming an alpha level of 0.05, a statistical power of 0.80, and a small to medium effect size (f = 0.2). Based on the fact that the current protocol has a therapist check-in component, a sample size recruitment target of n = 220 was set to allow for sample attrition, thus estimating a drop-out rate of approximately 30%.

Recruitment Possible participants are approached through ads on a social network. Those interested in using the application are asked to access the study's website and follow the standard recruitment procedure. They are subsequently contacted via a telephone call, at which point the enrollment procedure is described.

Assignment to study group The participants are randomly assigned to one of the three trial arms, using the software Randomizer.org. Randomization is performed by a research assistant using a simple (unrestricted) randomization sequence that assigns three unique numbers per participant; the number assigned is either 1, 2, or 3 according to the number of the experimental conditions. To conceal the allocation mechanism, the same research assistant will monitor the assessments and allow access to the application for the participants in the waitlist control group, after 6 weeks. The principal investigator and the statisticians running the data analysis will remain blinded to the study condition until the completion of the study.

Monitoring study implementation. Three clinical psychologists, members of the study team, screen for the risk of unintended effects or harm to the participants (i.e., clinically significant increase in depressive symptomatology, as measured by the CESD-R). The psychologists also monitor the weekly online evaluations and clinically interpret the CESD-R score of every participant. If the participant does not complete the CESD-R evaluation, a telephonic contact follows. If necessary, the supervisor can decide to interrupt the participant's access to the application and make a further referral.

ELIGIBILITY:
Inclusion Criteria:

* Romanian-speaking adults (18 years or older)
* Access to a computer, a smartphone (Android or iOS) and Internet
* A PHQ-9 score between 10 and 16

Exclusion Criteria:

* Undergoing treatment - medication and/or psychotherapy
* Substance abuse problems
* Psychotic symptoms
* Organic brain disorders (e.g., dementia)
* Self-injury or harming others
* Serious legal or health issues that would prevent from using the app
* Reporting scores larger than 1 to Question 9 (suicidal ideation) on the (PHQ-9)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 158 (Actual)
Dates: Start 2017-02-17 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Center for Epidemiologic Studies Depression Scale-Revised (CESD-R) (change from baseline) | Baseline, 1 week after baseline, 2 weeks after baseline, 3 weeks after baseline, 4 weeks after baseline, 5 weeks after baseline, post-intervention (6 weeks after baseline), Follow-up (3 months post-intervention)
  The CESD-R is a 20-item self-report instrument, which measures symptoms of depression in nine different groups: sadness (dysphoria), loss of interest (anhedonia), appetite, sleep, thinking/concentration, guilt (worthlessness), tired (fatigue), movement (agitation), and suicidal ideation. Participants rate each item on a five-point Likert scale, from 0 (not at all or less than one day) to 4 (nearly every day for 2 weeks) and refer to a time frame of a week or so. The Total CESD-R Score is calculated as a sum of responses to all 20 questions. The CESD-R exhibited good psychometric properties, including high internal consistency, strong factor loadings, and theoretically consistent convergent and divergent validity with anxiety, schizotypy, and positive and negative affect. CESD-R has been used previously on the Romanian population and was found to have adequate psychometric properties.

SECONDARY OUTCOMES:
The Positive and Negative Affect Scale (PANAS) (change from baseline) | Baseline, mid-intervention (3 weeks after baseline), post-intervention (6 weeks after baseline), Follow-up (3 months after post-intervention)
  The Positive and Negative Affect Scale (PANAS) is a 20-item self-report questionnaire designed to assess mood. It consists of 10 items that address positive affect (PA) and 10 items that address negative affect (NA). Participants rate each item on a five-point Likert scale, from 1 (very slightly/not at all) to 5 (extremely). The PANAS can be used to assess mood on various time scales by altering the instructions. For the purposes of this study a two-week timeframe has been used. The validity and internal consistency of the PANAS are good, with test-retest reliability being the highest for the "general" temporal instruction. The PANAS has been used previously on the Romanian population and was found to have adequate psychometric properties.
The Behavioural Activation for Depression Scale - Short Form (BADS-SF)(change from baseline) | Baseline, mid-intervention (3 weeks after baseline), post-intervention (6 weeks after baseline), Follow-up (3 months after post-intervention)
  The Behavioural Activation for Depression Scale - Short Form (BADS-SF) is an instrument designed to be administered weekly to measure changes in avoidance and activation over the course of the Behavioral Activation (BA) treatment for depression. The BADS consists of 9 items grouped into two subscales (Activation and Avoidance/Rumination). Respondents rate each item on a seven-point Likert scale ranging from 0 (not at all) to 6 (completely). The scale enjoys good psychometric properties. BADS-SF has been used previously on the Romanian population and was found to have adequate psychometric properties.
Satisfaction with Life (SWL) (change from baseline) | Baseline, mid-intervention (3 weeks after baseline), post-intervention (6 weeks after baseline), Follow-up (3 months after post-intervention)
  Satisfaction with Life (SWL) is a five-item scale designed to measure global cognitive judgments of one's life satisfaction. Participants rate each of the 5 items using a seven-point scale that ranges from 7 (strongly agree) to 1 (strongly disagree). The SWL has been shown to be a valid and reliable measure of life satisfaction, which can be used with a wide range of age groups. SWL has been used previously on the Romanian population and was found to have adequate psychometric properties.

OTHER OUTCOMES:
The Dysfunctional Attitudes Scale Short Form (DAS-SF) (change from baseline) | Baseline, mid-intervention (3 weeks after baseline), post-intervention (6 weeks after baseline), Follow-up (3 months after post-intervention)
  DAS was designed to measure the intensity of dysfunctional attitudes that, according to the cognitive theory of depression, contribute to vulnerability for depression. For the purpose of this study, the short form of this scale was used. The Dysfunctional Attitudes Scale-Short Form (DAS-SF) consists of two subscales: "dependency" (6 items) and "perfectionism/performance evaluation" (11 items). The 17 items are rated on a seven-point Likert scale, from 1 (total disagreement) to 7 (total agreement). DAS-SF possesses good psychometric properties in terms of model fit, reliability and convergent construct validity. DAS-SF has been used previously on the Romanian population and was found to have adequate psychometric properties.
The Beliefs Scale (BS) (change from baseline) | Baseline, mid-intervention (3 weeks after baseline), post-intervention (6 weeks after baseline), Follow-up (3 months after post-intervention)
  The Beliefs Scale (BS) measures irrational beliefs. It consists of 20 items and responders indicate the level of agreement/disagreement with each item using a five-point Likert scale that ranges from 1 (strongly disagree) to 5 (strongly agree). The BS shows good psychometric properties regarding construct and discriminant validity. This scale has been used previously on the Romanian population and was found to have adequate psychometric properties.
The Automatic Thoughts Questionnaire (ATQ) (change from baseline) | Baseline, mid-intervention (3 weeks after baseline), post-intervention (6 weeks after baseline), Follow-up (3 months after post-intervention)
  he Automatic Thoughts Questionnaire (ATQ) is a 15-item self-report measure used to assess depression-related cognitions. Participants rate, on a five-point Likert scale from 1 (never) to 5 (almost all the time), the frequency of a given thought over the past week. A higher score shows a higher frequency of automatic thoughts. The psychometric properties of the ATQ have been adequately demonstrated in previous studies. The ATQ has been successfully used on the Romanian population before.
Satisfaction with the Application Scale | Mid-intervention (3 weeks after baseline), post-intervention (6 weeks after baseline)
  Satisfaction with the Application Scale consists of 10 items that assess users' satisfaction with the application, its difficulty level, attractiveness, and subjective utility. The first 8 items are rated on a three-point scale, ranging from 0 to 2. Each response scale is personalized to the content of the item (e.g., How attractive did you find the exercises included in the application? - 0 = rather unattractive, 1 = attractive enough; 2 = very attractive). Item 9 assesses the application globally, with the participant being asked to give an overall grade between 1 (minimum) and 10 (maximum). Item 10 asks the participants if they would recommend the application to a friend ("yes" or "no" answer). This scale has been used previously by the same research team, in a study investigating the same mobile phone app.
The Application Use Scale | 1 week after baseline, 2 weeks after baseline, 3 weeks after baseline, 4 weeks after baseline, 5 weeks after baseline, post-intervention (6 weeks after baseline)
  The Application Use Scale consists of 8 items that assess weekly quantitative app usage aspects: the effort invested in homework (1 item), number of practiced exercises (1 item), number of read courses (1 item), frequency of general application use (1 item), and frequency of every exercise use (4 items). This scale has been used previously by the same research team, in a study investigating the same mobile phone app.

CONTACTS AND LOCATIONS:
Overall Officials: Cezar Giosan, PhD, Principal Investigator — Babeș-Bolyai University
Locations (1):
- Babeș-Bolyai University, Cluj-Napoca, Cluj, Romania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Giosan C, Cobeanu O, Mogoase C, Szentagotai A, Muresan V, Boian R. Reducing depressive symptomatology with a smartphone app: study protocol for a randomized, placebo-controlled trial. Trials. 2017 May 12;18(1):215. doi: 10.1186/s13063-017-1960-1. PMID 28494802
- See also: Study description and recruitment link — http://binedispus.ro